CLINICAL TRIAL: NCT04961307
Title: Evaluation of Heart Function in Breast Cancer Patients Using Trastuzumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cardiac safety study
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Cardiotoxicity; Antitumor Drugs; Breast Cancer; Trastuzumab
Keywords: Cardiac safety; Antitumor drugs; Breast Cancer; Trastuzumab
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with breast cancer using trastuzumab
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — 30 female breast cancer patients using trastuzumab, collected demographic and clinical information of all patients before chemotherapy, performed echocardiography (conventional echocardiography, three-dimensional spot tracking technology), and collected blood samples to detect plasma biology Markers (TnT, BNP, GDF-15, topoisomerase

SUMMARY:
By dynamically observing the changes of echocardiogram and biomarkers in breast cancer patients using trastuzumab, evaluate the effect of trastuzumab on cardiac function; determine the sensitivity of echocardiography and biomarker indicators And specificity, explore effective and specific early warning indicators, and provide technical support for the evaluation of the cardiac safety of anti-tumor drugs.

DETAILED DESCRIPTION:
Thirty female breast cancer patients using trastuzumab, collected demographic and clinical information of all patients before chemotherapy, performed echocardiography (conventional echocardiography, three-dimensional spot tracking technology), and collected blood samples to detect plasma biology Markers (TnT, BNP, GDF-15, topoisomerase), follow-up echocardiography and biomarkers at 1 month, 3 months and 6 months after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer (18-70 years old)
* Patients who are planning to undergo trastuzumab for the first time

Exclusion Criteria:

* Organic heart disease such as coronary heart disease, heart valve disease, cardiomyopathy
* liver and kidney failure
* severe cerebrovascular disease
* chronic obstructive pulmonary disease
* rheumatic immune system disease
* other tumors

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 30 female breast cancer patients using trastuzumab, collected demographic and clinical information of all patients before chemotherapy, performed echocardiography (conventional echocardiography, three-dimensional spot tracking technology), and collected blood samples to detect plasma biology Markers (TnT, BNP, GDF-15, topoisomerase)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Time ending | 6 months
  180 days after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided